CLINICAL TRIAL: NCT06002984
Title: Effectiveness of Intraoperative Neuromonitoring to Identify and Preserve External Branch of Superior Laryngeal Nerve During Thyroid Surgery
Brief Title: Effectiveness of Intraoperative Neuromonitoring of External Branch of Superior Laryngeal Nerve in Thyroid Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su-jin Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2303-075-1411
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Laryngeal Nerve Injuries; Thyroidectomy; Voice Change
Keywords: External branch of the superior Laryngeal Nerve
MeSH Terms: conditions — Laryngeal Nerve Injuries; Dysphonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Using neuromonitoring to find EBSLN (Experimental): With neuromonitoring of the EBSLN using nerve monitoring system Intervention Device: Neuromonitoring to find EBSLN
  Interventions: Device: Using Neuromonitoring to find EBSLN
- No using neuromonitoring to find EBSLN (No Intervention): Without neuromonitoring of the EBSLN using nerve monitoring system

INTERVENTIONS:
Device: Using Neuromonitoring to find EBSLN — intraoperative neuromonitoring to preserving external branch of superior laryngeal nerve during thyroid surgery
  Arms: Using neuromonitoring to find EBSLN

SUMMARY:
The frequent occurrence of impaired function in the external branch of the superior laryngeal nerves following thyroid surgery is recognized as a prevalent complication leading to a diminished quality of life. The objective of this randomized controlled trial (RCT) is to assess the efficacy of neuromonitoring during thyroid surgery in order to safeguard the integrity of these nerves.

DETAILED DESCRIPTION:
With increased interest in quality of life after thyroidectomy, preservation of proper vocal cord function and voice quality is an important issue in thyroid surgery. External branch of the superior laryngeal nerve (EBSLN) and recurrent laryngeal nerve (RLN) are crucial organs for innervation and integration of laryngeal muscular system. The EBSLN innervates the cricothyroid muscle (CTM), which is important in adjusting the tension and length of the vocal cords. Damage of the EBSLN leads to CTM dysfunction, resulting in difficulty with high pitch phonation and decreased pitch range and reduced voice projection, which are important for voice professionals. As the intraoperative neuromonitoring was utilized as an adjunctive and objective tool to confirm the nerve presence and integrity, application of the intraoperative neuromonitoring system to confirm EBSLN function pre- and post-dissection of the upper thyroid pole can be regarded as an effective method to preserve cricothyroid muscle function. However, it remains unclear whether there is any intraoperative neuromonitoring techniques-added value to the clinical outcome of thyroidectomy in terms of identification of EBSLN and preserved voice performance. Therefore, this study could provide strong evidence of the application of the intraoperative neuromonitoring during thyroid surgery to identify and preserve EBSLN function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo thyroid surgery
* Patients who understand and agree to take part in this study

Exclusion Criteria:

* If the thyroid tumor is suspected to invade adjacent organs (esophagus, trachea, carotid artery, jugular vein etc.)
* Patients who are required with lateral compartment neck dissection
* Patients with recurrent thyroid cancer
* Patients with palsy of recurrent laryngeal nerve or superior laryngeal nerve external branch in the past or present
* Patients with a history of vocal cord and larynx disease
* History of hyperthyroidism (e.g., Graves' disease)
* Taking anticoagulants (aspirin, warfarin, etc.) before surgery
* Disorders of coagulation
* In the case of women, pregnant women and breastfeeding patients
* Patients judged inappropriate by clinical trial researcher

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification rate of EBSLN | during operation
  Visual identification rate, Electrostimulatory identification rate

SECONDARY OUTCOMES:
Change of results about questionnaire for quality of voice | up to postoperative 1 month, 3 months and 6 months
  Voice Handicap Index-10 [0~40], higher scores mean worse voice disorder
Changes of Vocal outcome | up to postoperative 1 month, 3 months and 6 months
  Visual Analogue Scales (VAS) [0~100%], 0% = no voice, full disability ; 100% = normal voice
Measurements of Vocal function | up to postoperative 1 month, 3 months and 6 months
  Maximum Phonation Time (MPT)
Vocal evaluation | up to postoperative 1 month, 3 months and 6 months
  GRBAS (Grade, Rough, Breathy, Asthenia, and Strain)
Changes of Vocal fold vibration patterns | up to postoperative 1 month, 3 months and 6 months
  EGG (electroglottography) assessment of voice
Changes of Vocal outcome by Computerized Acoustic Analysis | up to postoperative 1 month, 3 months and 6 months
  Multi-Dimensional Voice Program (MDVP)
Changes of Voice Pitch | up to postoperative 1 month, 3 months and 6 months
  Real-time pitch (RTP)

CONTACTS AND LOCATIONS:
Overall Officials: Su-Jin Kim, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SJ, Lee KE, Oh BM, Oh EM, Bae DS, Choi JY, Myong JP, Youn YK. Intraoperative neuromonitoring of the external branch of the superior laryngeal nerve during robotic thyroid surgery: a preliminary prospective study. Ann Surg Treat Res. 2015 Nov;89(5):233-9. doi: 10.4174/astr.2015.89.5.233. Epub 2015 Oct 28. PMID 26576402
- [Background] Kim JI, Kim SJ, Xu Z, Kwak J, Ahn JH, Yu HW, Chai YJ, Choi JY, Lee KE. Efficacy of Intraoperative Neuromonitoring in Reoperation for Recurrent Thyroid Cancer Patients. Endocrinol Metab (Seoul). 2020 Dec;35(4):918-924. doi: 10.3803/EnM.2020.778. Epub 2020 Dec 23. PMID 33397044
- [Background] Potenza AS, Phelan EA, Cernea CR, Slough CM, Kamani DV, Darr A, Zurakowski D, Randolph GW. Normative intra-operative electrophysiologic waveform analysis of superior laryngeal nerve external branch and recurrent laryngeal nerve in patients undergoing thyroid surgery. World J Surg. 2013 Oct;37(10):2336-42. doi: 10.1007/s00268-013-2148-9. PMID 23838931
- [Background] Barczynski M, Konturek A, Stopa M, Honowska A, Nowak W. Randomized controlled trial of visualization versus neuromonitoring of the external branch of the superior laryngeal nerve during thyroidectomy. World J Surg. 2012 Jun;36(6):1340-7. doi: 10.1007/s00268-012-1547-7. PMID 22402975
- [Background] Jonas J, Bahr R. Neuromonitoring of the external branch of the superior laryngeal nerve during thyroid surgery. Am J Surg. 2000 Mar;179(3):234-6. doi: 10.1016/s0002-9610(00)00308-1. PMID 10827327
- [Background] Babinska D, Barczynski M, Oseka T, Sledzinski M, Lachinski AJ. Comparison of perioperative stress in patients undergoing thyroid surgery with and without neuromonitoring-a pilot study. Langenbecks Arch Surg. 2017 Jun;402(4):719-725. doi: 10.1007/s00423-016-1457-5. Epub 2016 Jun 14. PMID 27299585
- [Background] Cirocchi R, Arezzo A, D'Andrea V, Abraha I, Popivanov GI, Avenia N, Gerardi C, Henry BM, Randolph J, Barczynski M. Intraoperative neuromonitoring versus visual nerve identification for prevention of recurrent laryngeal nerve injury in adults undergoing thyroid surgery. Cochrane Database Syst Rev. 2019 Jan 19;1(1):CD012483. doi: 10.1002/14651858.CD012483.pub2. PMID 30659577
- [Background] Dionigi G, Boni L, Rovera F, Bacuzzi A, Dionigi R. Neuromonitoring and video-assisted thyroidectomy: a prospective, randomized case-control evaluation. Surg Endosc. 2009 May;23(5):996-1003. doi: 10.1007/s00464-008-0098-3. Epub 2008 Sep 21. PMID 18806939
- [Background] Lifante JC, McGill J, Murry T, Aviv JE, Inabnet WB 3rd. A prospective, randomized trial of nerve monitoring of the external branch of the superior laryngeal nerve during thyroidectomy under local/regional anesthesia and IV sedation. Surgery. 2009 Dec;146(6):1167-73. doi: 10.1016/j.surg.2009.09.023. PMID 19958945